CLINICAL TRIAL: NCT04718688
Title: Exploring the Use of the Cognitive Orientation to Daily Occupational Performance Approach (CO-OP) With Children With Executive Functions Deficits Following Severe Acquired Brain Injury: a Single Case Experimental Design Study
Brief Title: Exploring the Use of the CO-OP With Children With EF Functions Deficits Following ABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M2 COOP_HL
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Acquired Brain Injury
Keywords: Cognitive Orientation to daily Occupational Performance; Rehabilitation; Executive functions; child acquired brain injury; occupational performance
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: single case experimental study design (SCED) with multiple baselines across individuals and behaviors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CO-OP intervention (Experimental): CO-OP intervention
  Interventions: Other: CO-OP rehabilitation

INTERVENTIONS:
Other: CO-OP rehabilitation — The intervention was included within the child's conventional rehabilitation program.
  In the CO-OP original protocol, the child sets 3 goals. Here, we concentrated on two rather than three goals, as addressing three occupations per session seemed too ambitious given the children's cognitive profile (the third goal served as control goal).
  We chose to increase the number of sessions to 14 (two sessions per week for seven weeks, vs ten in the original protocol).
  The global strategy was taught to the child at the first session. The following sessions consisted of an iterative process of implementation of the global strategy in the context of guided discovery to identify domain specific strategies to overcome performance ''breakdowns" the children were experiencing when performing the self-selected tasks. In addition, "homework" was assigned to encourage the application and practice. Parents were invited to attend the sessions if it was possible for them.

SUMMARY:
Purpose:

Acquired brain injury (ABI) in childhood are the cause of disabling motor, cognitive and behavioural disorders, with severe consequences on the later development of autonomy and learning, with long-term repercussions on independence for activities of daily living, and social and professional integration. Among cognitive disorders, executive function (EF) deficits are among the most frequent and disabling, with major consequences on the development of autonomy and the course of schooling and learning. The Cognitive Orientation to daily Occupational Performance (CO-OP) could be an interesting approach for the rehabilitation of these consequences. CO-OP is a performance-based treatment approach for children and adults who experience difficulties performing the skills they want to, need to or are expected to perform. CO-OP is a specifically tailored, active client-centered approach that engages the individual at the meta-cognitive level to solve performance problems. Focused on enabling success, the CO-OP approach employs collaborative goal setting, dynamic performance analysis, cognitive strategy use, guided discovery, and enabling principles. It has been shown to be effective in a variety of populations, but has been little explored in children with ABI.

Objectives To assess whether the use of CO-OP could be of interest in children with executive functions deficits following ABI, to improve their occupational performance, their executive functioning in everyday life and their cognitive processes constituting EF.

DETAILED DESCRIPTION:
Method

* Single case experimental study with multiple baselines across individuals and behaviors
* 14 individual sessions of CO-OP intervention.
* Two goals trained, one control goal.
* Different assessments used : Canadian Occupational Performance Measure (COPM), the Goal Attainment Scales (GAS), the Children's Cooking Task (CCT) and parent- and teacher-ratings of the Behavior Rating Inventory of Executive Functions (BRIEF) questionnaire.

ELIGIBILITY:
Inclusion criteria were:

* Age 8 to 14 years
* Diagnosis of ABI, sustained at least 6 months previously, still attending an in- or outpatient rehabilitation program following injury
* Evidence of a dysexecutive syndrome on the neuropsychological assessment
* Normal vision and hearing (with appropriate correction if necessary)
* Sufficient language skills to understand and to communicate explicitly

Exclusion criteria were:

* Non-French-speaking child or parents
* Sensory-motor or visual impairments precluding participation in the study
* Intellectual deficit (Full-Scale Intellectual Quotient (IQ)<70), or severe impairments in comprehension, memory or attention, incompatible with understanding and choosing rehabilitation goals and participating in 45-minutes sessions
* Neurological, psychiatric, genetic or learning disability diagnosed prior to the ABI
* Severe anxiety or depression symptoms

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Goal Attainment Scaling (GAS) change | Baseline to 3-months post-intervention (Three times per week during baseline and intervention phase for each 3 chosen-goal ; one time at 3-months post-intervention)
  Goal Attainment Scaling (GAS) is a method for writing personalized evaluation scales in order to quantify progress toward defined goals.
  GAS methodology consists in:
  * Defining a rehabilitation goal;
  * Choosing an observable behaviour that reflects the degree of goal attainment;
  * Defining the patient's initial level with respect to the goal;
  * Defining five goal attainment levels (ranging from a ''no change'' to a ''much better than expected outcome'');
  * Evaluating the patient after a defined time interval;
  * Calculating the overall attainment score for all the rehabilitation goals. A five-point scale is used: ''-2'' is the initial pretreatment (baseline) level, ''-1'' represents progression towards the goal without goal attainment, ''0'' is the expected level after treatment, (and therefore, the ''most likely'' level after treatment), ''+1'' represents a better outcome than expected, and ''+2'' is the best possible outcome that could have been expected for this goal.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Before baseline, at immediate post-intervention, at 3-months post-intervention.
  This semi-structured interview helps children/parents identify problematic occupations in different daily areas. COPM will be used: (1) To determine (only with the child) the 4 problematic occupations identified as the most important (3 will be used as target goals, while the 4 will serve as a control goal); (2) To determine changes in occupational performance in self-selected goals: children and parents will rated their performance and satisfaction associated with these 4 occupations. Performance and satisfaction are rated by children and parents on a scale of 1 to 10 (1= not at all able to perform the activity (performance) / not at all satisfied with the way the activity is performed (satisfaction); 10 = perfectly able to perform the activity (performance) / perfectly satisfied with the way the activity is performed (satisfaction). A difference of 2 points between pre- and post-intervention is clinically significant.
Behavior Rating Inventory of Executive Function (BRIEF) | Three times during baseline, at immediate post-intervention, at 1- and 3-months post-intervention
  The parent and teacher report forms of the Behavior Rating Inventory of Executive Function (BRIEF, or BRIEF-A for adults'version) provide an ecological assessment of executive functioning through its repercussions in family and school context. Currently, this questionnaire is the best validated and most widely used in children in various congenital, developmental or acquired conditions. The outcome measure is the Global Executive Composite score (GEC) T-Scores (Mean: 50; SD: 10; clinical range cutoff: T-Scores≥65).
Children's cooking task | pre-intervention, immediate post-intervention and 3-months post-intervention
  The Children's Cooking Task (CCT) is an ecological standardized task designed to assess EF during actual execution of a complex task: the child is asked to prepare a chocolate cake and a fruit cocktail following two simple, highly structured, illustrated recipes with numbered steps. The CCT was used as a secondary outcome measure in this study in order to determine whether children transferred progress in problem-solving, acquired through strategies discovered with CO-OP, onto the performance of a complex task, unrelated to the trained goals.

CONTACTS AND LOCATIONS:
Overall Officials: Helene LEBRAULT, Mec, Principal Investigator — Hopitaux de Saint-Maurice
Locations (1):
- Saint Maurice Hospitals, Saint-Maurice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lebrault H, Chavanne C, Abada G, Latinovic B, Varillon S, Bertrand AF, Oudjedi E, Krasny-Pacini A, Chevignard M. Exploring the use of the Cognitive Orientation to daily Occupational Performance approach (CO-OP) with children with executive functions deficits after severe acquired brain injury: A single case experimental design study. Ann Phys Rehabil Med. 2021 Sep;64(5):101535. doi: 10.1016/j.rehab.2021.101535. Epub 2021 Jul 17. PMID 33933689